CLINICAL TRIAL: NCT01555671
Title: Is There Any Effect of Meperidine on the Length of Duration of Labor? A Prospective Randomized Controlled Trial.
Brief Title: Study of the Effectiveness of Administration of Meperidine on the Length of Active Phase of Labor in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Orhan SAHIN, M.D., MD,, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 02-11-11-Rev-1
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Labor Pain
Keywords: labor,; meperidine,; active phase,; duration of labor
MeSH Terms: conditions — Labor Pain | interventions — Meperidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized parallel double blind plasebo controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both drug provider and patient do not know which drug or placebo was given
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- meperidine administration group (Active Comparator): Infusion bags were prepared and labelled as Bag A (meperidine group), containing 25 mg meperidine (Aldolan; Liba Laboratuarları, Istanbul, Turkey) .Providers and patients were blinded to the contents of the bags until the conclusion of the study. Meperidine or placebo were administered by intravenous infusion by means of injectors containing 0.5ml of solution.
  Interventions: Drug: Meperidine
- plasebo group (Placebo Comparator): Bag B (placebo group), containing 0.5ml of normal saline solution. Providers and patients were blinded to the contents of the bags until the conclusion of the study.Meperidine or placebo were administered by intravenous infusion by means of injectors containing 0.5ml of solution.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Meperidine — 0.5 ml meperidine injection intravenously injected in randomly selected patients
  Other Names: Aldolan 100 mg/2 ml
  Arms: meperidine administration group
Drug: Saline — 0.5 ml saline solution injection intravenously injected in randomly selected patients
  Other Names: 0.90% w/v of NaCl
  Arms: plasebo group

SUMMARY:
This study aims to evaluate the effect of meperidine on the length of active phase of labor in nulliparous or multiparous women, who will be randomized into two (control and study) groups. Our hypothesis is that the use of meperidine during active labor has no effect on the duration of labor.

DETAILED DESCRIPTION:
* Our aim is to examine the effect of the opioid derivative meperidine used during labor on the duration of labor in singleton pregnancies.
* The sample size was calculated using the Number Cruncher Statistical System (NCSS) / PASS 2007. Power 80% and significance level (α) 0.05, the mean (mean) ± standard deviation (SD) of the first 20 individuals included in the control group of the study (296.04 ± 170.02) and has minimal clinical significance for the active phase of labor from previous studies. We found that the sample size should be 200 (100/100) considering the duration (30 minutes).
* A Simple randomisation using a random-number table was performed by the independent nurse staff, who took no further part in the study.Using the sealed envelope technique, parturients were randomly allocated to two groups: A meperidine group and B normal saline group
* Age, height, weight, body mass index (BMI), gravida, parity, week of gestation, expected fetal weight (EFW), hemoglobin (Hb) and hematocrit (Hct) values and episiotomy requirements were recorded in two groups.Gender, birth weight, 1st and 5th minute Apgar scores and presence of meconium aspiration of the newborns in two groups were recorded.
* During labor, oxytocin induction was not performed during the latent phase in accordance with the routine protocol of our hospital. Pregnant women in both groups were given oxytocin (Synpitan® amp) at a concentration of 1% by 10 drops/min by performing amniotomy when Bishop score was 6 or cervix dilation was 4 cm and when 70% effacement was achieved. In the meperidine group, when the cervical opening was 6 cm and 70% washout, 25 mg iv bolus injection of meperidine (2.5 ml) was administered. The same amount (2.5 ml) of physiological saline was administered intravenously to the subjects in the control group. The patients were followed in NST until 10 cm clearance and 100% effacement. This time was recorded as active phase time. The time from the end of the active phase period to the birth of the baby was recorded as the duration of the second phase of birth.
* The primary outcome of interest in this study is the duration of active phase of labor .

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 38 and 42 weeks
* live fetus
* cephalic presentation
* in active phase of labour

Exclusion Criteria:

* placenta previa, placental abruption
* caesarean section or any uterine scarring
* multiple gestation
* fetal macrosomia (≥4000 g)
* meperidine allergy
* use any kind of labour induction or augmentation before on admission for delivery in our hospital

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2015-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orhan SAHIN, MD, Study Director — Ministery of Health
Locations (1):
- Prof.Dr.Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Leong WL, Sng BL, Sia AT. A comparison between remifentanil and meperidine for labor analgesia: a systematic review. Anesth Analg. 2011 Oct;113(4):818-25. doi: 10.1213/ANE.0b013e3182289fe9. Epub 2011 Sep 2. PMID 21890889
- [Result] Sica-Blanco Y, Rozada H, Remedio MR. Effect of meperidine on uterine contractility during pregnancy and prelabor. Am J Obstet Gynecol. 1967 Apr 15;97(8):1096-100. doi: 10.1016/0002-9378(67)90471-1. No abstract available. PMID 6021289
- [Result] Sosa CG, Balaguer E, Alonso JG, Panizza R, Laborde A, Berrondo C. Meperidine for dystocia during the first stage of labor: A randomized controlled trial. Am J Obstet Gynecol. 2004 Oct;191(4):1212-8. doi: 10.1016/j.ajog.2004.03.017. PMID 15507943
- [Result] Sosa CG, Buekens P, Hughes JM, Balaguer E, Sotero G, Panizza R, Piriz H, Alonso JG. Effect of pethidine administered during the first stage of labor on the acid-base status at birth. Eur J Obstet Gynecol Reprod Biol. 2006 Dec;129(2):135-9. doi: 10.1016/j.ejogrb.2005.11.033. Epub 2006 Jan 6. PMID 16406273
- See also: meperidine,duration of labor,induction of labor — http://www.nlm.nih.gov/medlineplus/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to be carried out between January 2012 and May 2012 in Kanuni Sultan Süleyman training and research hospital(Istanbul-Turkey), gynecology and obstetrics department.
Pre-assignment Details: A total of 449 patients were included in the study. 199 patients who did not meet the inclusion criteria were excluded from the study. The remaining 250 patients were randomized to the groups.
Groups:
- Study Group: Infusion bags were prepared and labelled as Bag A (meperidine group), containing 25 mg meperidine,0.5ml (Aldolan; Liba Laboratuarları, Istanbul, Turkey) .
- Control Group: Bag B (placebo group), containing 0.5ml of normal saline solution.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 125 | 125
Completed | 105 | 100
Not Completed | 20 | 25
Not completed — Physician Decision | 20 | 25

BASELINE CHARACTERISTICS:
Population: term pregnancies with active labor
Groups:
- Study Group: 0.5 ml meperidine injection intravenously injected in randomly selected patients
- Plasebo Group: 0.5 ml saline solution injection intravenously injected in randomly selected patients
- Total: Total of all reporting groups
Arm/Group | Study Group | Plasebo Group | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 125 | 250
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Of the 250 patients included in the study, 45 patients with cesarean indication were excluded from the study and baseline measurements were made on the remaining patient population.
  years
    number analyzed (Participants) | 105 | 100 | 205
    (all) | 25.21 (5.17) | 26.03 (4.8) | 25.83 (5.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 125 | 250
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: The Duration of Active Phase of Labour
Description: The primary outcome is to evaluate whether meperidine is effective in shortening the duration of the active phase of labor
Time Frame: 24h
Population: women giving birth at term period
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Meperidine Administration Group | Plasebo Group
Number analyzed (Participants) | 105 | 100
minutes | 249 (122) | 304 (167)
Statistical Analysis 1: Comparison: Meperidine Administration Group vs Plasebo Group; Test type: Other; p = 0.029, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 30

2. Secondary Outcome: Total Duration of Labour
Description: Total time of delivery of patients who gave birth including the second stage of delivery
Time Frame: 24h
Population: Total time of delivery of patients who gave birth including the second stage of delivery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Meperidine Administration Group | Plasebo Group
Number analyzed (Participants) | 105 | 100
minutes | 273 (129) | 331 (177)

3. Secondary Outcome: Duration of the Second Stage of Labour
Description: The period of time until the birth of the baby, since the patient being followed for delivery
Time Frame: 24h
Population: duration of the second stage of labour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Meperidine Administration Group | Plasebo Group
Number analyzed (Participants) | 105 | 100
minutes | 24 (15) | 27 (22)

ADVERSE EVENTS:
Time Frame: 24h
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/100
Other Adverse Events (participants affected / at risk) | 20/105 | 4/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=105) | Control Group (N=100)
emezis (Gastrointestinal disorders) | 20 (24) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No